CLINICAL TRIAL: NCT03988179
Title: Registration of Attentional Function as a Predictor of Incident Delirium
Brief Title: Predicting Delirium by Attentional Dysfunction
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, W ten Hoope, Prof. dr. W.A. van Gool, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL47720.018.014
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Delirium in Old Age
Keywords: Attention; Attentional dysfunction; Delirium; Preoperative
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Cholinesterase Inhibitor Prognosticator (ChIP) application for iPad — The first part of this application will be used, consisting of a visual vigilance test based on the Continuous Performance Test (CPT). Stimuli consist of a one digit number presented in the middle of the screen. For each trial the application randomly selects a specific number as the target stimulus. Patients are instructed to keep their dominant trigger finger close to the screen and press a button which is located at the bottom of the screen, whenever the target appears. In case another stimulus appears the patient is instructed to do nothing. Each stimulus is presented until the patient presses the button (maximum 3 sec.). Stimuli are presented in a random fashion with a 1, 2, 3, 4, or 5 second inter-stimuli-interval blank, which randomly varies. After an 8 stimuli practice trial, the test starts and a total of 50 stimuli are presented with a 50% target rate. Full-trial duration is approximately 5 minutes. During the trial, reaction time and accuracy of response are registered.

SUMMARY:
Rationale: Delirium is a common complication that occurs in various medical conditions. Validated models predicting delirium in individual patients are scarce and existing models tend to focus on demographic characteristics and comorbid conditions exclusively. Previous research has suggested that impairment of attentional function might serve as an early and specific individual predictor of incident delirium. Utilization of a test measuring attentional function in a clinically easy-to-use tool could potentially yield a pathophysiological monitor to identify individual patients at risk of evolving delirium and target future prophylactic treatment.

Objective: To assess the difference in preoperative intra-individual reaction time variability between postoperative delirium and non-delirium elderly non-dementia patients undergoing elective surgery. Study design: An observational prospective cohort study.

Study population: Elderly patients (70 years or older) undergoing elective surgery.

Main study parameters/endpoints: Preoperative intra-individual reaction time variability among postoperative non-delirium and delirium patients.

DETAILED DESCRIPTION:
Delirium is a common complication that occurs in various medical conditions. Development of delirium during admission is associated with an increase in length of hospital stay, complication rates, mortality and consequently higher healthcare expenditures. Besides these short-term consequences, delirium is detrimental to long-term outcome with an ensuing higher risk of dementia, institutionalization and death.

Development of delirium is associated with increasing age. The risk for postoperative delirium among elderly patients ranges from 4%-53%. Incidence differs between different surgical procedures and between emergency or elective surgery. A systematic review comparing general to regional anaesthetic procedures did not show significant differences in the risk for developing postoperative delirium.

Although an array of risk factors associated with development of delirium has been identified in numerous studies, validated models predicting delirium in individual patients are scarce.

Moreover, existing models tend to focus on demographic characteristics and comorbid conditions exclusively. Models predicting development of delirium by using individual pathophysiological markers involved in the evolution of delirium are absent.

Previous research has suggested that impairment of attentional function might serve as an early and specific individual predictor of incident delirium, even in previously cognitively undisturbed patients. So far only one study has prospectively assessed preoperative intra-individual reaction time variability as a predictor of postoperative delirium. This study was limited to elderly (age 70 years or older) patients undergoing elective hip and knee replacement and did not examine confounding factors such as preoperative use of (anti-cholinergic) drugs, preoperative presence of symptoms of depression, cognitive decline or impairment in activities of daily living making. Although this study showed significant higher preoperative intra-individual reaction time variability among patients developing postoperative delirium, no attempts to reproduce these findings in other surgical populations have been published to date, limiting external validity and practical implementation of these observations.

The investigators hypothesize that preoperative intra-individual reaction-time variability is an independent predictor of postoperative delirium. In this study the investigators aim at assessing the potential of preoperative administration of a short test of attentional function in predicting postoperative delirium in a population of elderly non-dementia patients undergoing major elective surgery. Utilization of a test measuring attentional function in a clinically easy-to-use tool could potentially yield a pathophysiological monitor to preoperatively identify individual patients undergoing elective surgery who are at an increased risk of evolving delirium and create a target for future prophylactic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Elective surgery involving thoracotomy, major abdominal surgery (e.g. esophageal, gastric, hepatic, pancreatic, colorectal resection by either laparotomy or laparoscopic approach), major pelvic surgery (e.g. radical cystectomy, radical hysterectomy), or major orthopedic surgery (e.g. knee or hip replacement)

Exclusion Criteria:

* Preceding diagnosis of dementia or Clinical Dementia Rating (CDR) scale of 1 or more
* Language barrier enough to hamper informed consent and iPad instructions
* Serious functional disability of the dominant hand (e.g. palsy, amputation, arthrodesis)

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly non-dementia patients undergoing major elective surgery.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-23 (Actual)

PRIMARY OUTCOMES:
Preoperative intra-individual reaction time variability. | 02-2014 / 06-2015
  To assess the difference in preoperative intra-individual reaction time variability between postoperative delirium and non-delirium elderly non-dementia patients undergoing elective surgery.

SECONDARY OUTCOMES:
Preoperative individual accuracy of reaction time response. | 02-2014 / 06-2015
  To assess the difference in preoperative accuracy of response on a reaction time test between postoperative delirium and non-delirium elderly non-dementia patients undergoing elective surgery.
Association between intra-individual reaction time variability on the ChIP application for iPad and development of delirium, defined as a positive score on the CAM on any given moment during the first 5 days postoperatively. | 02-2014 / 06-2015
  For each subject preoperative intra-individual reaction time variability will be determined using the standard deviation (SD) of individual preoperative reaction times (continuous variable). To determine the association between preoperative intra-individual reaction time variability and development of postoperative delirium odds ratios (OR) along with 95% confidence intervals (CI) will be calculated using multivariate logistic regression. A cut-off will be made at 1 SD above total group mean average for scores on intra-individual reaction time. Presence of delirium will be defined as a positive score on the CAM on any given moment during the first 5 days postoperatively.
Association between accuracy of reaction time response on the ChIP application for iPad and delirium, defined as a positive score on the CAM on any given moment during the first 5 days postoperatively. | 02-2014 / 06-2015
  For each subject preoperative individual accuracy of reaction time response will be determined by the total of target stimuli missed (continuous variable). To determine the association between individual accuracy of response and development of postoperative delirium odds ratios (OR) along with 95% confidence intervals (CI) will be calculated using multivariate logistic regression. A cut-off will be made at 1 SD above total group mean average for scores on individual accuracy of response. Presence of delirium will be defined as a positive score on the CAM on any given moment during the first 5 days postoperatively.
Sensitivity and specificity of a combined index of preoperative intra-individual reaction time variability and accuracy of response in predicting delirium. | 02-2014 / 06-2015
  To determine the sensitivity and specificity of a combined index of preoperative reaction time variability and accuracy of response in predicting postoperative delirium among elderly non-dementia patients undergoing elective surgery.

CONTACTS AND LOCATIONS:
Overall Officials: W. A. van Gool, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Undecided